CLINICAL TRIAL: NCT00812838
Title: The Efficacy of Botulinum Toxin Type a in Treating Peyronie's Disease
Brief Title: H-22411: BOTOX® for Peyronie's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mohit Khera (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Mohit Khera, Assistant Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-07-40-04
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Peyronie's Disease
MeSH Terms: conditions — Penile Induration | interventions — Botulinum Toxins, Type A; Crossing Over, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 units of Botulinum Toxin Type A (Experimental): Injection solution will consist of 100 units of BOTOX® in 10 cc of preservative free normal saline
  Interventions: Drug: 100 units of Botulinum Toxin Type A
- Normal saline (Placebo Comparator): Injection solution will consist of 10 cc preservative free normal saline
  Subjects had the choice of crossing over to ARM 1 at the end of 16 weeks.
  Cross-over: For subjects in Arm 2, crossover to BOTOX treatment will begin after the Week 16 Visit by repeating the study schedule as for Week 0 to Week 16.
  Interventions: Other: Preservative free normal saline; Drug: 100 units Botulinum Toxin A

INTERVENTIONS:
Drug: 100 units of Botulinum Toxin Type A — Approximately 20 to 30 injections of 100 units of BOTOX® given with a 20 gage needle directly into the penile plaque
  Other Names: BOTOX®
  Arms: 100 units of Botulinum Toxin Type A
Other: Preservative free normal saline — Approximately 20 to 30 injections of 10cc of preservative free normal saline given with a 20 gage needle directly into the penile plaque
  Arms: Normal saline
Drug: 100 units Botulinum Toxin A — Approximately 20 to 30 injections of 100 units of BOTOX® given with a 20 gage needle directly into the penile plaque
  Other Names: Cross-over
  Arms: Normal saline

SUMMARY:
Peyronie's disease is a condition in which a plaque, or hard lump, forms on the penis. It causes hardened tissue, pain, and an abnormal bending in the penis. These symptoms are more severe during an erection. Significant bending of the penis can result in pain, poor erections, and an inability to engage in sexual intercourse.

This disease affects about 3% of the male population. The average age of onset of this disease is 57 years old. The cause of the disease is unknown. However, many believe that it may be due to trauma to the penis (such as injury or extremely vigorous sexual activity).

DETAILED DESCRIPTION:
Treatments for this disease have been limited and often unsuccessful. The goal of treatment is to reduce pain and maintain sexual function. Oral medicines that prevent plaque formation and promote plaque breakdown have not been effective. Many patients with the disease will require injections of medicines directly into the plaque. These injections have been used for over 50 years in the treatment of major Peyronie's disease. The disease often resolves on its own without treatment. Surgery may be performed to remove hardened tissue in the penis. However, surgery is not done during the first 12 months of the disease.

There are 2 phases of the disease: the active phase and the inactive phase. The active phase usually occurs during the first 12 months of the disease. The stabilization of the plaque is known as the inactive phase. We are inviting men with stable disease to take part in this study which will test BOTOX® versus a placebo (a placebo contains no medicine).

This will be a randomized, placebo-controlled, cross-over, single-center trial. The placebo group has the option to cross over to the treatment arm (ARM 1) of the study at the end of their 16 weeks of placebo arm (ARM 2). Study drug is Botulinum toxin type A (BOTOX®). Subjects who meet the inclusion criteria for the study will be randomized to either the treatment or placebo arm.

* Treatment: Injection solution will consist of 100 units of BOTOX® in 10 cc of preservative free normal saline, or
* Placebo: Injection solution will consist of 10 cc preservative free normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stable Peyronie's plaques.
* Males at least 18 years of age
* Must give informed consent.

Exclusion Criteria:

* Subjects in the active phase of Peyronie's disease.
* Subjects with less than 1 year history of Peyronie's disease.
* Subjects taking oral medications for Peyronie's disease which include Trental, Viagra, vitamin E, colchicines, L-arginine, and tamoxifen. There will be a 2 week wash-out period if patients are on these medications.
* Subjects with more than 1 penile plaque will be excluded from the study.
* Subjects with calcified plaques demonstrated by ultrasound will be excluded from the study.
* Known allergy or sensitivity to any components of the study medication (botulinum toxin A), anesthetics, or any other product associated with the treatment and general study procedures.
* Any medical condition or neuromuscular disorder that may put the patient at increased risk with exposure to botulinum toxin A (BTX-A), including myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis.
* Patient taking aminoglycosides or any drug known to interfere with neuromuscular transmission.
* Patient has hemophilia or other clotting factor deficiencies or disorders that cause bleeding diathesis.
* Patient must not be taking aspirin, non-steroidal anti-inflammatory drugs, or Coumadin for 7 or more days prior to Botox injection.
* Episode of unstable angina pectoris, myocardial infarction, transient ischemic attack, or cerebrovascular accident within the past 6 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08-07 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Khera, MD, MBA, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published in aggregate.

REFERENCES:
- [Background] Khera M, Boone TB, Smith CP. Botulinum toxin type A: a novel approach to the treatment of recurrent urethral strictures. J Urol. 2004 Aug;172(2):574-5. doi: 10.1097/01.ju.0000130652.27541.22. No abstract available. PMID 15247734

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: 100 units of Botulinum Toxin Type A Injection solution will consist of 100 units of BOTOX® in 10 cc of preservative free normal saline
- Placebo Comparator: Normal saline Injection solution will consist of 10 cc preservative free normal saline.
  Optional Cross-over: For subjects in Arm 2, crossover to BOTOX treatment will begin after the Week 16 Visit by repeating the study schedule as for Week 0 to Week 16.
Period: Treatment Period of 16 Weeks
Arm/Group | Experimental | Placebo Comparator
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Optional Crossover of 16 Weeks
Arm/Group | Experimental | Placebo Comparator
Started (Optional crossover did not apply to the experimental arm (ARM 1)) | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per the study protocol, two arms of the study are analyzed; the experimental arm and the placebo arm
  *4 subjects cross over from ARM 2 to ARM 1after 16 weeks. Crossover subjects were added to Experimental Group for analysis with Adverse Events, International Index of Erectile Function, Penile Curvature, and Reduction in Plaque Size*
Groups:
- Experimental: 100 units of Botulinum Toxin Type A Injection solution will consist of 100 units of BOTOX® in 10 cc of preservative free normal saline
  *Crossover subjects were added to Experimental Group for analysis*
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo Comparator | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants] — Population: Per the study protocol, two arms of the study are analyzed; the experimental arm and the placebo arm
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 6 | 12
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per the study protocol, two arms of the study are analyzed; the experimental arm and the placebo arm
  years | 58.86 (4.741) | 57.83 (3.710) | 58.38 (4.154)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Per the study protocol, two arms of the study are analyzed; the experimental arm and the placebo arm
  Participants
    Female | 0 | 0 | 0
    Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per the study protocol, two arms of the study are analyzed; the experimental arm and the placebo arm
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 6 | 6 | 12
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per the study protocol, two arms of the study are analyzed; the experimental arm and the placebo arm
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 6 | 5 | 11
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Average Percent Change of Penile Curvature in Degrees
Description: Measured by a protractor from pictures taken at baseline (pre-treatment screening visit) and end of treatment at week 16
  *Crossover subjects were added to Experimental Group for analysis*
  Negative value equates to a reduction in curvature Positive value equates to an increase in curvature
Time Frame: Baseline (Pre-Treatment Screening Visit) to end of treatment at week 16
Population: *Crossover subjects were added to Experimental Group for analysis*
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Placebo Comparator: Normal saline Injection solution will consist of 10 cc preservative free normal saline
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 10 | 6
percent change | -21.73 (57.69) | 2.429 (81.59)
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; Test type: Superiority; p = 0.5154, t-test, 2 sided — This will be a pilot study; it was assessed that 10 subjects in each arm, for a total of 20 subjects, will allow us to determine if the therapy is effective. To allow for screen failures, 45 subjects are planned for screening

2. Secondary Outcome: Change in Penile Blood Flow for Peak Systolic Velocity (PSV) and End-diastolic Velocity (EDV)
Description: Results of penile doppler ultrasound from baseline/screening visit to end of treatment at week 16 will be compared.
  peak systolic velocity (PSV) and end-diastolic velocity (EDV) are assessed here.
  Change is calculated as week 16 values - screening visit values
  Negative values are a decrease in velocity Positive values are an increase in velocity
Time Frame: Baseline (Pre-Treatment Screening Visit) to end of treatment at week 16
Population: *Penile Doppler ultrasound was not performed on optional crossover patients. Data reflects scores derived from Experimental and Placebo group analysis.
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Normal Saline: Injection solution will consist of 10 cc preservative free normal saline
  Preservative free normal saline: Approximately 20 to 30 injections of 10cc of preservative free normal saline given with a 20 gage needle directly into the penile plaque
Arm/Group | 100 Units of Botulinum Toxin Type A | Normal Saline
Number analyzed (Participants) | 6 | 6
cm/s
  Pre injection Right PSV | -0.65670 (5.505) | -9.0170 (11.43)
  Pre injection Right EDV | -2.10200 (6.798) | -0.8667 (3.771)
  Pre injection Left PSV | -1.263 (9.032) | -6.4330 (12.04)
  Pre injection Left EDV | -10.27 (8.261) | -6.75 (11.63)
  5 minutes right PSV | 5.185 (28.48) | 2.1330 (6.425)
  5 minutes right EDV | -11.05 (19.56) | -0.1417 (3.944)
  5 minutes left psv | 2.863 (17.68) | -6.6830 (22.76)
  5 minutes left edv | -2.4 (10.80) | 3.5 (10.16)
  15 minutes right PSV | 6.917 (20.91) | -15.52 (34.44)
  15 minutes right EDV | -10.22 (22.82) | 1.55 (5.001)
  15 minutes left PSV | 7.183 (10.81) | -15.10 (40.93)
  15 minutes left EDV | -2.267 (11.58) | 3.367 (6.046)
Statistical Analysis 1: Comparison: 100 Units of Botulinum Toxin Type A vs Normal Saline; This will be a pilot study; it was assessed that 10 subjects in each arm, for a total of 20 subjects, will allow us to determine if the therapy is effective. To allow for screen failures, 45 subjects are planned for screening. This analysis pertains to both categories; Test type: Superiority; p = 0.3009, t-test, 2 sided — This applies to 100 units of Botulinum Toxin Type A arm vs the Normal saline arm

3. Secondary Outcome: Change in Penile Blood Flow for Diameter
Description: Results of penile doppler ultrasound from the baseline/screening visit to end of treatment at week 16 will be compared.
  Diameter is assessed here.
  Change is calculated as week 16 values - screening visit values
  Negative values are a decrease in diameter Positive values are an increase in diameter
Time Frame: Baseline (Pre-Treatment Screening Visit) to end of treatment at week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 6 | 6
cm
  Pre injection right Diameter | -0.29 (0.8539) | 0.1700 (0.7208)
  Pre injection left diameter | 0.04167 (0.5869) | 0.3983 (0.4565)
  5 minute right diameter | 1.34200 (4.006) | 0.2917 (0.6719)
  5 minute left diameter | -0.75330 (2.551) | 0.0750 (0.9000)
  15 minute right diameter | -1.43700 (3.952) | -0.3550 (0.6469)
  15 minute left diameter | -0.43500 (2.571) | -0.1867 (1.203)
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; This will be a pilot study; it was assessed that 10 subjects in each arm, for a total of 20 subjects, will allow us to determine if the therapy is effective. To allow for screen failures, 45 subjects are planned for screening; Test type: Superiority; p = 0.0166, t-test, 2 sided — This applies to 100 units of Botulinum Toxin Type A arm vs the Normal saline arm

4. Secondary Outcome: Change in Penile Plaque Size
Description: Results of ultrasound at baseline/screening visit to end of treatment at week 16 will be compared.
  *Crossover subjects were added to Experimental Group for analysis*
  Change is calculated as week 16 values values minus screening visit values
  Increase in value equates to increased plaque size Decrease in value equates to decreased plaque size
Time Frame: Baseline (Pre-Treatment Screening Visit) to end of treatment at week 16
Population: *Crossover subjects were added to Experimental Group for analysis*
Measure: Mean (Standard Deviation); unit: cubic millimeters
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 10 | 6
cubic millimeters
  screening visit | 717.5 (827.4) | 485.8 (599.6)
  week 16 | 198.9 (220.8) | 319.0 (252.2)
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = .8566, t-test, 2 sided — Threshold for statistical significance was <0.05

5. Secondary Outcome: Changes in International Index of Erectile Function Scores (IIEF)
Description: Subject's average scores on IIEF at baseline/screening visit to end of treatment at week 16 are compared
  The subscale measures self-reported erectile function. Maximum score is 30, Minimum is 0. A score of 0 is the absolute best outcome. A score of 30 is the absolute worst outcome. Erectile Function score is a summation of questions 1,2,3,4, and 15. This study is assessing their erectile function and not the other subscales.
  The other subscale scores are :
  1. Orgasmic Function (Questions 9, 10); Maximum score = 10, Minimum score = 0
  2. Sexual Desire (Questions 11, 12); Maximum score = 10, Minimum score = 0
  3. Intercourse Satisfaction (Questions 6, 7, 8); Maximum score = 15, Minimum score = 0
  4. Overall Satisfaction (Question 13, 14): Maximum score = 10, Minimum score = 0
  Subscales are not combined to make a total composite score.
  *Crossover subjects were added to Experimental Group for analysis*
Time Frame: Baseline (Pre-Treatment Screening Visit) to end of treatment at week 16
Population: *Crossover subjects were added to Experimental Group for analysis*
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Placebo Comparator
Number analyzed (Participants) | 10 | 6
score on a scale
  Screening Visit | 15.60 (11.75) | 21 (12.13)
  Week 16 | 17.20 (11.61) | 21.50 (11.74)
Statistical Analysis 1: Comparison: Experimental vs Placebo Comparator; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0286, t-test, 2 sided — Threshold for statistical significance is <0.05

ADVERSE EVENTS:
Time Frame: 2 years, 8 months
Arm/Group | 100 Units of Botulinum Toxin Type A | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 5/10 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 Units of Botulinum Toxin Type A (N=10) | Normal Saline (N=6)
Cold (Immune system disorders) | 2 (2) | 0 (0) — Cold - no treatment provided
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — No treatment was provided
Bruising (Vascular disorders) | 2 (2) | 0 (0) — No treatment was provided
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — No treatment was provided
small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — 1, small bowel obstruction; pain pressure in his abdomen
seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — seasonal allergies
increased frequent urination (Renal and urinary disorders) | 1 (1) | 0 (0) — increased frequent urination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT00812838/Prot_SAP_000.pdf